CLINICAL TRIAL: NCT02384005
Title: The Feasibility of Self or Partner-assisted Digital Anal Exam Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Alan G Nyitray, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HSC-SPH-13-0671; 1R21CA181901-01A1 (NIH)
Record Dates: First submitted 2015-03-03; First posted 2015-03-10 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Anus Neoplasms
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Self-anal exam arm (Other): Study only has one arm.
  Interventions: Other: Self-anal exam arm

INTERVENTIONS:
Other: Self-anal exam arm — After a short pre-test the clinician will use a model to show a normal and diseased anal canal and then use pictures to show a self-DAE. The clinician will describe how to do a self-DAE for single men and partners. Next, the clinician will ask the participant to lower his pants for collection of anal human papillomavirus (HPV) DNA and cytology. The clinician will conduct a DAE and then participants will do self-DAE done in private. Then the research assistant will demonstrate the computer-assisted self-interview. When participants return to the clinician to receive the DAE results, the clinician will conduct a safety-related interview. The clinician will treat external anal disease, triage internal anal disease, and ask to be notified if a participant has any anus-related concerns in the following week. A complete appointment will require 70 minutes for singles and 105 minutes for couples. The PI will later conduct 3 focus groups.

SUMMARY:
There is no standard screening protocol for anal cancer even as disease incidence increases. This single-visit study will clarify if single persons can do a self-digital anal exam, or perhaps the exam requires a partner, or if, in fact, the exam requires a clinician for reasons of safety, accuracy, or acceptability.

The investigators hypothesize that men having sex with men's digital anal exam (DAE) findings will have moderate or substantial agreement with a nurse practitioner DAE for detecting an anal abnormality (defined as condylomas, hemorrhoids, fissures, and malignant tumors). As a secondary hypothesis the investigator believe a partner-assisted DAE conducted within a couple will have better agreement with the nurse practitioner DAE than will a self-DAE conducted by a single person.

DETAILED DESCRIPTION:
There is no standard screening protocol for anal cancer even as disease incidence and mortality increases; however, a digital anorectal exam (also called a digital rectal exam) will play a role in any recommended protocol. Critically, fewer digital anorectal exams are being performed by physicians even though it is a simple and quick procedure. If men who have sex with men (MSM) can learn to examine the anal canal, then detection and treatment of early cancers among this population may increase. This single-visit Phase II feasibility study will investigate increasing digital anal exam (DAE) use to enhance screening for anal cancer among MSM aged 27-80 years. The investigators hypothesize that MSM's DAE findings will have moderate or substantial agreement with a nurse practitioner DAE for detecting an anal abnormality (defined as condylomas, hemorrhoids, fissures, and malignant tumors). As a secondary hypothesis the investigators believe a partner-assisted DAE conducted within a couple will have better agreement with the nurse practitioner DAE than will a self-DAE conducted by a single person. It is not proposed that lay persons recognize specific conditions but, rather, that any abnormality should trigger a doctor visit. The specific aims are:

1. Estimate the agreement between the digital anal exams of 200 MSM and the gold standard of a highly experienced nurse practitioner during a single clinical visit.

   This aim will answer the question: under optimal circumstances, will MSM report accurate findings after performing their own DAE?
2. Determine factors independently associated with concordance of MSM and nurse practitioner DAEs including age, single men vs. men in couples, race, ethnicity and waist circumference.

   This aim will provide insight into which MSM are more likely to perform accurate DAEs.
3. Assess DAE acceptability, self-efficacy, safety, and intentions-to-seek subsequent care.

This aim will answer the question: will lay-performed DAEs have sufficient acceptability and safety and trigger appropriate follow-up care?

The goal is to advance knowledge of how to increase use of digital anal exams to reduce anal cancer morbidity and mortality. The study will clarify if single persons can do a self-digital anal exam, or perhaps the exam requires a partner, or if, in fact, the exam requires a clinician for reasons of safety, accuracy, or acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Men who are aged 27-80 years
* Acknowledge sex with men in their lifetime
* Reside in Harris County, Texas
* Understand and speak English.

Exclusion Criteria:

* Current doctor's diagnosis of anal condyloma, hemorrhoids, fissures, or anal cancer

Ages: 27 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Kappa agreement will be calculated between lay person and nurse practitioner on the anal exam results. | This cross-sectional design measures agreement on Day 1.

SECONDARY OUTCOMES:
Odds ratios will be calculated for the association between partnership status and concordance between participant and clinician. | This cross-sectional design collects data for the odds ratios on Day 1
Odds ratios will be calculated for the association between age and concordance between participant and clinician. | This cross-sectional design collects data for the odds ratios on Day 1
Odds ratios will be calculated for the association between waist circumference and concordance between participant and clinician. | This cross-sectional design collects data for the odds ratios on Day 1
Odds ratios will be calculated for the association between race and concordance between participant and clinician. | This cross-sectional design collects data for the odds ratios on Day 1
Odds ratios will be calculated for the association between ethnicity and concordance between participant and clinician. | This cross-sectional design collects data for the odds ratios on Day 1
Number of persons who state that a self-DAE is an acceptable procedure. | This cross-sectional design collects these data on Day 1
Number of persons with adverse events after conducting a self-DAE. | This cross-sectional design collects these data on Day 1
Number of persons who state they have the ability to conduct a self-DAE. | This cross-sectional design collects these data on Day 1
Number of persons who state they intend to seek subsequent care in the event of an abnormal result to a self-DAE. | This cross-sectional design collects these data on Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Alan G. Nyitray, PhD, Principal Investigator — University of Texas School of Public Health at Houston
Locations (1):
- University of Texas School of Public Health, Houston, Texas, United States

REFERENCES:
- [Derived] Nyitray AG, Hicks JT, Hwang LY, Baraniuk S, White M, Millas S, Onwuka N, Zhang X, Brown EL, Ross MW, Chiao EY. A phase II clinical study to assess the feasibility of self and partner anal examinations to detect anal canal abnormalities including anal cancer. Sex Transm Infect. 2018 Mar;94(2):124-130. doi: 10.1136/sextrans-2017-053283. Epub 2017 Aug 23. PMID 28835533